CLINICAL TRIAL: NCT04694417
Title: Prevention of Leg Cramps Using Compression Stockings or Magnesium Supplements in the Age Group of 50 to 84: a Study Protocol for a Randomised Controlled Trial
Brief Title: Prevention of Leg Cramps Using Compression Stockings or Magnesium Supplements in the Age Group of 50 to 84
Acronym: CramP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tampere University Hospital (Other)
Collaborators: Tampere University (Other)
Responsible Party: Principal Investigator, Tuomas-Heikki Koskela, Professor (tenure track), Tampere University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: TampereUH99
Record Dates: First submitted 2020-12-30; First posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Muscle Cramp; Stockings, Compression; Magnesium
MeSH Terms: conditions — Muscle Cramp | interventions — Stockings, Compression; Magnesium

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The participants assigned to the two tablet groups will be blinded to the intervention. The magnesium and placebo tablets that are used in the trial will be identical in terms of packaging and appearance. The compression stocking group cannot be blinded, but the participants will not know their allotted intervention until they have received it by mail delivery. The statisticians will be blinded to the group allocation by using codes to label the three groups and will randomly assign outcome assessors to the follow-up. The allocation sequence will be concealed until the end of the study. The allocation code will be stored in a separate file.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Compression stocking (Experimental): Compression stockings are mainly used for the prevention and reduction of lower limb oedema or venous thrombosis. There are three compression classes used in health care. The compression stocking group of the study will receive CE-marked stockings within the compression class of 1 (25-40 mmHg compression). The correct size for the compression stockings will be defined by the reported circumference of the participant's ankle and calf. The participants will be given instructions to put the stockings on immediately after getting out of bed in the morning and to take them off before going to bed in the evening for the last four weeks of the study. Stockings within the mild compression class have no harmful effects on individuals when the exclusion criteria are considered. The participants will be instructed to communicate with a dedicated research assistant via e-mail or phone in case of any problems or questions.
  Interventions: Other: Compression stocking
- Magnesium (Active Comparator): Magnesium is a mineral substance which regulates many biochemical reactions in the body, for example protein synthesis and the function of the muscles and nerves. It has a significant role in controlling blood sugar, blood pressure, energy generation and the formation of the bones. The recommended dietary allowance for magnesium is 420 mg for males and 320 mg for females over 50 years old. Dark green vegetables, leguminous plants, nuts, seeds and wholegrains are good sources of magnesium (11,12).
  In the average Finnish diet, the recommendation is usually exceeded, and excessive amounts of magnesium in the body are extremely rare. The magnesium arm of the study will take oral tablets containing 620 mg of magnesium hydrochloride daily for the last four weeks of the study, which is equivalent to 250 mg of pure magnesium per day. The magnesium tablets for this study were manufactured and analysed by the Pharmia pharmaceutical company in Finland.
  Interventions: Dietary Supplement: Magnesium tablet
- Placebo (Placebo Comparator): The placebo tablets will consist of microcrystalline cellulose, magnesium stearate (anti-caking agent) and silicon dioxide. The placebo tablets were manufactured and analysed by the Pharmia pharmaceutical company in Finland. The placebo arm will receive placebo tablets to be taken daily for the last four weeks of the study. The participants will not know whether they are randomised into the magnesium arm or the placebo arm. The packaging and the appearance of the placebo and magnesium tablets are identical.
  Interventions: Other: Placebo tablet

INTERVENTIONS:
Other: Compression stocking — Please see the description of the intervention in another section
  Arms: Compression stocking
Dietary Supplement: Magnesium tablet — Please see the description of the intervention in another section
  Arms: Magnesium
Other: Placebo tablet — Please see the description of the intervention in another section
  Arms: Placebo

SUMMARY:
Leg cramps are painful sensations of tightening in the muscles of the legs, that are often associated with secondary insomnia. They are common especially at an older age. There is no evidence that any method of prevention of nocturnal leg cramps would be both safe and effective. There are no previous trials concerning cramp prevention by using compression stockings. The objective of this study is to assess in a prospective randomised controlled trial whether leg cramps can be prevented by daily use of knee-length compression stockings or magnesium supplements.

DETAILED DESCRIPTION:
Leg cramps are painful sensations of tightening in the muscles of the legs that commonly appear during the night and are often associated with secondary insomnia. They are common especially in older age. There is no evidence that any method of prevention of nocturnal leg cramps is both safe and effective. There are no previous trials concerning cramp prevention by using compression stockings. The objective of this study is to assess in a prospective randomised controlled trial whether leg cramps can be prevented by the daily use of knee-length compression stockings or magnesium supplements.

Methods The study will be set in Finland, and 50-84-year-old volunteers will be recruited through Google Ads, the Finnish Health Library and Finnish primary health care centres. The participants must have a minimum of two episodes of leg cramps per week for the past four weeks to be included in the study. The participants (n = 225) will be allocated to three equal groups: the compression stocking arm, the magnesium supplement arm and the placebo arm. The participants will go through four weeks of follow-up without intervention, and then another four weeks of follow-up with the assigned intervention. The material for the study will be collected through electronic questionnaires.

Discussion This protocol describes a study that compares compression stockings, magnesium supplements and placebo for the prevention of leg cramps. The results of this study can significantly improve knowledge on the methods of preventing leg cramps.

ELIGIBILITY:
Inclusion Criteria:

* Minimum of two leg cramps per week in the past four weeks.
* Age from 50 to 84 years.

Exclusion Criteria:

* Peripheral artery disease (confirmed or suspected).
* Peripheral artery bypass surgery.
* Grave peripheral neuropathy or any sensory disorder.
* Allergy to the material of the compression stockings.
* Grave renal failure (GFR under 30 ml/min).
* The use of a magnesium carbonate product (e.g. Rennie® or Berocca®).
* Cardiac failure with pulmonary oedema or massive lower limb swelling.
* Lower limb soft tissue problems, including skin transplant, thinned skin, varicose ulcer, necrosis and any infection.
* Lower limb deformity or atypical shape or size that could prevent the usage of compression stockings.
* Continuous usage of compression stockings for any other reason than leg cramps.

Ages: 50 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
The change in quantity of leg cramps | 8 weeks
  The change in quantity of leg cramps from the four-week follow-up period (prior to the intervention) to the four-week intervention period will be assessed on the basis of the participants' responses to the survey. The number of cramps will be recoded on a weekly online survey during four weeks before intervention and during the four-week intervention period. The change in the number of cramps from the four-week period prior the intervention to the intervention period will be calculated. The difference between groups will be analyzed by one-way analysis of variance of repeated measurements.

SECONDARY OUTCOMES:
The change in intensity of leg cramps | 8 weeks
  The possible change in the intensity of leg cramps from the four-week follow-up period (prior to the intervention) to the four-week intervention period will be assessed on the basis of the participants' responses to the survey. The intensity of cramps will be recoded on a weekly online survey during the four weeks before intervention and during the four-week intervention period. The possible change in the intensity of cramps from the four-week period prior the intervention to the intervention period will be assessed.
The change in quantity of nocturnal awakening due to the cramps | 8 weeks
  The change in the quantity of nocturnal awakenings due to the cramps from the four-week follow-up period (prior to the intervention) to the four-week intervention period will be assessed on the basis of the participants' responses to the survey. The number of cramps will be recoded on a weekly online survey during four weeks before intervention and during the four-week intervention period. The change in the number of nocturnal awakenings due to the cramps from the four-week period prior the intervention to the intervention period will be calculated. The difference between groups will be analyzed by one-way analysis of variance of repeated measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Tuomas Koskela, Docent, Study Director — Tampere University Hospital

IPD SHARING:
Plan to Share IPD: No
The full protocol will be available in open access format. The datasets generated and analysed during this trial will be available from the corresponding author on reasonable request.

REFERENCES:
- [Derived] Joensuu J, Mustajoki PP, Mustonen PK, Kaila M, Koskela T. Prevention of leg cramps by using compression stockings or magnesium supplements in the 50-84 age group: study protocol for a randomised controlled trial. Trials. 2021 Nov 29;22(1):860. doi: 10.1186/s13063-021-05753-0. PMID 34844641